CLINICAL TRIAL: NCT07019571
Title: Evaluating the Impact of Transcranial Direct Current Stimulation on Urge in Body-Focused Repetitive Behaviors
Brief Title: tDCS and Urge in BFRBs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gopalkumar Rakesh (Other)
Responsible Party: Sponsor-Investigator, Gopalkumar Rakesh, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 101505
Record Dates: First submitted 2025-05-23; First posted 2025-06-13 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Repetitive Compulsive Behavior
Keywords: picking; biting; transcranial stimulation
MeSH Terms: conditions — Bites and Stings | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- active multifocal Transcranial Direct Current Stimulation (tDCS) (Experimental): participants receive 13-min of active multifocal tDCS targeting the left dorsolateral prefrontal cortex. tDCS will be delivered offline for 13 minutes (1.5mA, 10 seconds ramp in/out).
  Interventions: Device: Wireless Multichannel Transcranial Current Stimulator (tDCS); Behavioral: Cue exposure; Behavioral: Boredom induction
- sham multifocal Transcranial Direct Current Stimulation (tDCS) (Sham Comparator): Sham stimulation will be identical to active but electrical current will only be ramped in/out at the beginning and end of the 13-min period.
  Interventions: Device: Wireless Multichannel Transcranial Current Stimulator (tDCS); Behavioral: Cue exposure; Behavioral: Boredom induction

INTERVENTIONS:
Device: Wireless Multichannel Transcranial Current Stimulator (tDCS) — tDCS will be delivered for 13 minutes (active) or only at the beginning and end of the 13 minute period (sham) using Neuroelectrics Instrument Controller software and a battery-driven Starstim 8-channel transcranial direct current stimulator with 1cm2 ceramic electrodes and SIGNAGEL conductive saline gel.
Behavioral: Cue exposure — Participants will undergo three, twenty-second trials of exposure to individualized cues at the top of the established urge hierarchy, previously determined to precede picking or biting behaviors before and after tDCS.
Behavioral: Boredom induction — Participants will be left in the testing room without access to a cellphone or reading materials for 2 different 6 minute periods.

SUMMARY:
The goal of this study is to find out if brain stimulation can help people stop skin-picking or nail-biting. The study wants to answer two main questions:

1. Does brain stimulation reduce the urge to pick skin or bite nails after those urges are triggered?
2. Does brain stimulation reduce how often people pick their skin or bite their nails?

Participants will:

* Talk about their skin-picking, nail-biting, and other mental health concerns
* Be placed in situations that make them want to pick or bite
* Rate how strong their urges are before and after brain stimulation Researchers will compare real brain stimulation to a placebo (a fake version that looks the same but has no effect) to see if the real stimulation works to reduce skin-picking and nail-biting urges and behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent (as established by clinical interview), and voluntary, signed informed consent prior to the performance of any study specific
* Ability and willingness to perform study-relevant clinical assessments and tDCS
* Endorses mild to extreme intensity of urges to pick or bite their skin or nails

Exclusion Criteria:

* Any unstable medical, psychiatric, or neurological condition (including active or otherwise problematic suicidality) that may necessitate urgent treatment
* Daily use of psychotropic medications that substantially lower seizure threshold (e.g., clozapine)
* History of psychosis, mania, major neurological disorder, significant head trauma, or seizures/epilepsy
* Current suicidal intent
* Any major neurological disease or history of major head trauma, including concussion with extended loss of consciousness, or of psychosurgery
* Current or suspected pregnancy
* Endorsing possible contraindications for tDCS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in subjective urge | baseline and post intervention, approximately 90 minutes
  Individuals will rate their urge to pick using a scale (1-10) with a higher score meaning greater urge. They will rate their urge three times in a row, at two different time-points.
Change in subjective distress | baseline and post intervention, approximately 90 minutes
  Individuals will rate their distress using a scale (1-10) with a higher score meaning greater distress. They will rate their distress three times in a row, at two different time-points.
Change in picking or biting behavioral frequency | baseline and post intervention (approximately 90 minutes)
  Picking or biting behaviors will be assessed via two 6-minute blocks of visual observation, before and after tDCS. The frequency of the behaviors observed will be collected in each block. Change in total frequency between blocks will be calculated.
Change in picking or biting behaviors duration | baseline and post intervention (approximately 90 minutes)
  Picking or biting behaviors will be assessed via two 6-minute blocks of visual observation, before and after tDCS. Duration of the behaviors observed will be collected in each block. Change in total duration between blocks will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Gopalkumar Rakesh, MD, Study Director — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No